CLINICAL TRIAL: NCT02453009
Title: CHemotherapy Plus Enzalutamide In First Line Therapy for Castration Resistant prOstate caNcer
Brief Title: Addition of Enzalutamide to First Line Docetaxel for Castration Resistant Prostate Cancer
Acronym: CHEIRON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santa Chiara Hospital (Other)
Responsible Party: Principal Investigator, Orazio Caffo, MD, Santa Chiara Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TN-CHEIRON
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Docetaxel 75 mg/m² intravenously on day 1 every 3 weeks for 8 cycles, plus oral prednisone 10 mg daily for 24 weeks plus oral enzalutamide 160 mg daily for 24 weeks
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Enzalutamide
- Arm B (Active Comparator): Docetaxel 75 mg/m² intravenously on day 1 every 3 weeks for 8 cycles, plus oral prednisone 10 mg daily for 24 weeks
  Interventions: Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel — Pharmaceutical form:solution Route of administration: intravenous
Drug: Prednisone — Pharmaceutical form:tablet Route of administration: oral
Drug: Enzalutamide — Pharmaceutical form : soft gelatin capsules Route of administration: oral
  Other Names: Xtandi
  Arms: Arm A

SUMMARY:
The aim of this study is to verify if the addition of enzalutamide to docetaxel is able to improve the disease control in first line CRPC patients.

DETAILED DESCRIPTION:
CHEIRON trial is a phase II randomized study comparing docetaxel plus enzalutamide to docetaxel alone as first line for castration resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-confirmed prostate adenocarcinoma.
2. Metastatic disease.
3. Progressive disease while receiving hormonal therapy or after surgical castration documented by at least one of the following:

   * Increase in measurable disease (RECIST 1.1) [15], and/or
   * Appearance of new lesions, including those on bone scan consistent with progressive prostate cancer, and/or
   * Rising PSA defined as 2 sequential increases above a previous lowest reference value. Each value must be obtained at least 1 week apart. A PSA value of at least 2 ng/ml is required at study entry.
   * Effective castration (serum testosterone levels ≤0.50 ng/dL) by orchiectomy and/or LHRH agonists or antagonist with or without anti-androgens.

     i. If the patient has been treated with LHRH agonists or antagonist (i.e., without orchiectomy), then this therapy should be continued.

   ii. If patients were either started on complete androgen blockade, or had a PSA response (defined by any reduction in PSA sustained for at least 3 months) after adding an antiandrogen, prior anti-androgen therapy should be stopped before randomization: at least 6 weeks for bicalutamide and nilutamide, and at least 4 weeks for flutamide, megestrol acetate and any other hormonal therapy.
4. More than 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status <2 (see Appendix 2).
6. Ability to fill the quality of life questionnaire
7. Patient compliance and geographic proximity that allow adequate follow-up.
8. Presence of signed and dated IRB-approved patient informed consent form prior to enrollment into the study.

Exclusion Criteria:

1. Prior chemotherapy for prostate cancer, except estramustine and except adjuvant/neoadjuvant treatment completed >3 years ago.
2. Prior treatment with abiraterone acetate and/or enzalutamide
3. Less than 28 days elapsed from prior treatment with estramustine, radiotherapy or surgery to the time of randomization. Patients may be on biphosphonates prior to study entry.
4. Prior isotope therapy, whole pelvic radiotherapy, or radiotherapy to >30% of bone marrow.
5. History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
6. History of seizure or any condition that may predispose to seizure (eg, prior cortical stroke or significant brain trauma). History of loss of consciousness or transient ischemic attack within 12 months of randomization;
7. Inadequate organ and bone marrow function
8. Contraindications to the use of corticosteroid treatment.
9. Clinically significant cardiovascular disease
10. Any of the following within 3 months prior to randomization: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event.
11. Hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene;
12. Prior malignancy. Adequately treated basal cell or squamous cell skin or superficial (pTis, pTa, and pT1) bladder cancer are allowed, as well as any other cancer for which chemotherapy has been completed >5 years ago and from which the patient has been disease-free for >5 years.
13. Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization.
14. Any other condition which in the judgment of the investigator would place the subject at undue risk or interfere with the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Rate of patients without progression (according to guideline of Prostate Cancer Clinical Trials Working Group 2 - PCWG2) | 6 months after docetaxel first administration
  Rate of patients without progression (according to guideline of Prostate Cancer

SECONDARY OUTCOMES:
Rate of objective response according to RECIST criteria | 6 months after docetaxel first administration
  Rate of objective response according to RECIST criteria
Rate of biochemical response according to PCWG2 | 6 months after docetaxel first administration
  Rate of biochemical response according to PCWG2
Kaplan-Meier estimates of progression-free survival | 6 months after docetaxel first administration
  Kaplan-Meier estimates of progression-free survival
Kaplan-Meier estimates of overall survival | 6 months after docetaxel first administration
  Kaplan-Meier estimates of overall survival
Kaplan-Meier estimates of biochemical progression-free survival | 6 months after docetaxel first administration
  Kaplan-Meier estimates of biochemical progression-free survival
Rate of treatment-related mortality | 6 months after docetaxel first administration
  Rate of treatment-related mortality
Rate of toxicity-related protocol withdrawal | 6 months after docetaxel first administration
  Rate of toxicity-related protocol withdrawal
Scales of brief pain inventory (BPI) | 6 months after docetaxel first administration
  Scales of brief pain inventory (BPI
Analgesic score | 6 months after docetaxel first administration
  Analgesic score
Functional scales and items of FACT - P questionnaire | 6 months after docetaxel first administration
  Functional scales and items of FACT - P questionnaire
Type and grade of any adverse reaction to treatment, according to CTC-AE v. 4.03 | 6 months after docetaxel first administration
  Type and grade of any adverse reaction to treatment, according to CTC-AE v. 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Orazio Caffo, MD, Study Chair — Santa Chiara Hospital
Locations (1):
- Santa Chiara Hospital, Trento, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Caffo O, Ortega C, Nole F, Gasparro D, Mucciarini C, Aieta M, Zagonel V, Iacovelli R, De Giorgi U, Facchini G, Veccia A, Palesandro E, Verri E, Buti S, Razzini G, Bozza G, Maruzzo M, Ciccarese C, Schepisi G, Rossetti S, Maines F, Kinspergher S, Fratino L, Ermacora P, Nicodemo M, Giordano M, Sartori D, Scapoli D, Sabbatini R, Lo Re G, Morelli F, D'Angelo A, Vittimberga I, Lippe P, Carrozza F, Messina C, Galli L, Valcamonico F, Porta C, Pappagallo G, Aglietta M. Docetaxel and prednisone with or without enzalutamide as first-line treatment in patients with metastatic castration-resistant prostate cancer: CHEIRON, a randomised phase II trial. Eur J Cancer. 2021 Sep;155:56-63. doi: 10.1016/j.ejca.2021.06.016. Epub 2021 Aug 3. PMID 34358777